CLINICAL TRIAL: NCT02913248
Title: Short and Long Term Alterations of Subgingival and Salivary Microbiota in Relation to Periodontal Treatment
Brief Title: Salivary Bacterial Profiles in Relation to Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Forsyth Institute (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Daniel Belstrøm, DDS, PhD, Assistant professor, University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UCPH_OI_001
Record Dates: First submitted 2016-09-20; First posted 2016-09-23 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Periodontitis
Keywords: periodontitis; saliva; bacteria
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Conventional periodontal treatment (Experimental): 35 subjects diagnosed with manifest periodontitis, which will all receive standardized treatment according to protocol. In brief, this treatment includes professional tooth cleaning and thorough instruction in self-performed oral hygiene procedures. Clinical registrations and collection of microbiological samples (subgingival and saliva) will performed at baseline and 2, 6 and 12 weeks after treatment.
  Interventions: Procedure: Conventional periodontal treatment

INTERVENTIONS:
Procedure: Conventional periodontal treatment — Non-surgical periodontal treatment including thorough instruction in self-performed oral hygiene

SUMMARY:
The purpose of the present investigation is to record and compare bacterial compositions in subgingival plaque samples and saliva samples in subjects receiving periodontal treatment. The hypothesis is that the composition of the salivary microbiota might reflect local bacterial alterations in relation to periodontal treatment.

DETAILED DESCRIPTION:
In this study we plan to enroll 35 subjects with manifest periodontitis, which will be treated according to national and international guidelines. Clinical registration and collection of subgingival plaque samples and saliva samples will be performed at baseline and 2, 6 and 12 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

- Manifest chronic periodontitis according to international classification

Exclusion Criteria:

* Other treatment requiring oral conditions
* Systemic antibiotics within the latest 6 months
* Systemic diseases and medications with known associations to periodontitis
* Pregnancy and breastfeeding

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10; Primary Completion 2017-01-02 (Actual); Study Completion 2017-01-02 (Actual)

PRIMARY OUTCOMES:
Changes in α-diversity in saliva samples collected . | Baseline and 12 weeks
  Comparison of α-diversity in saliva samples collected before periodontal treatment and 12 weeks after treatment

SECONDARY OUTCOMES:
Specis specific changes in saliva samples collected | Baseline and 12 weeks
  Comparison of relative abundance of bacterial species in saliva samples collected before periodontal treatment to samples collected 12 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Belstrøm, DDS, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Department of Odontology, Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data will be handled anonymously

REFERENCES:
- [Derived] Grande MA, Belstrom D, Damgaard C, Holmstrup P, Thangaraj SS, Nielsen CH, Palarasah Y. Complement split product C3c in saliva as biomarker for periodontitis and response to periodontal treatment. J Periodontal Res. 2021 Jan;56(1):27-33. doi: 10.1111/jre.12788. Epub 2020 Jul 18. PMID 32681659
- [Derived] Grande MA, Belstrom D, Damgaard C, Holmstrup P, Kononen E, Gursoy M, Gursoy UK. Salivary concentrations of macrophage activation-related chemokines are influenced by non-surgical periodontal treatment: a 12-week follow-up study. J Oral Microbiol. 2019 Dec 9;12(1):1694383. doi: 10.1080/20002297.2019.1694383. eCollection 2020. PMID 31893018